CLINICAL TRIAL: NCT06091540
Title: Pilot Randomized Controlled Trial on the Feasibility and Efficacy of Individual SH+ Intervention for Earthquake Survivors
Brief Title: Feasibility and Efficacy of Individual SH+ Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Ceren Acarturk, Principal investigator, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.292.IRB3.135
Record Dates: First submitted 2023-10-16; First posted 2023-10-19 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Grief Disorder, Prolonged
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to the conditions of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feasibility and Efficacy of Individual SH+ Intervention (Experimental): The first phase of the study involves executing a pilot randomized controlled trial (RCT) with an earthquake-adapted iteration of the SH+ intervention. This phase will introduce modifications to the traditional SH+ approach. Unlike the conventional SH+ manual, which includes audio elements and paired discussions centered around specific topics, the adapted version will omit the audio components. Instead, the intervention will be delivered directly by the psychologist on a one-on-one basis. Additionally, while the original SH+ format involves paired discussions within a group setting, this study will focus on individual sessions. The intervention aims to provide a more personalized approach, promoting a more individualized and humane dimension to the healing process.
  Interventions: Behavioral: Feasibility and Efficacy of Individual SH+ Intervention
- Treatment as Usual (No Intervention): Participants will undergo random assignment to either the treatment as usual (TAU) condition or the intervention condition. Upon completion of all measurements, the control condition will be given the opportunity to receive the intervention.

INTERVENTIONS:
Behavioral: Feasibility and Efficacy of Individual SH+ Intervention — The key parameter of interest will be the extent of psychological distress encountered by the participants. In addition, various secondary outcomes will also be evaluated, encompassing depression, anxiety, post-traumatic stress disorder (PTSD) symptoms, psychosocial well-being, and grief levels. The evaluation of the intervention's effectiveness on the sample of interest will hinge on the comparison of scores obtained during the pretest and posttest measurement phases.
  Arms: Feasibility and Efficacy of Individual SH+ Intervention

SUMMARY:
The central aim of this research is to execute a randomized controlled trial (RCT) to assess the impact and effectiveness of the individually-delivered SH+ intervention among earthquake survivors in Türkiye. The principal focus lies in investigating the potential benefits of the intervention. The key parameter of interest will be the extent of psychological distress encountered by the participants. In addition, various secondary outcomes will also be evaluated, encompassing depression, anxiety, post-traumatic stress disorder (PTSD) symptoms, psychosocial well-being, and grief levels. The evaluation of the intervention's effectiveness on the sample of interest will hinge on the comparison of scores obtained during the pretest and posttest measurement phases. It is hypothesized that scores will exhibit a decline following the participants' engagement with the SH+ program over the span of five weeks. Specifically, the hypothesis being tested posits that there will be a notable reduction in depression, anxiety, post-traumatic stress, psychological distress, psychosocial impairment, and grief scores during the post-assessment stage in contrast to the pre-assessment stage. It is expected that the experimental condition and the control condition will demonstrate significant differences in depression, anxiety, post-traumatic stress, psychosocial impairment, and grief scores. The primary outcome measure of psychological distress will show a statistically significant difference between the experimental and control groups at both the immediate posttest assessment and the 3-month follow-up assessment.

DETAILED DESCRIPTION:
On February 6 2023, Türkiye experienced two consecutive major earthquakes measuring 7.6 and 7.8 on the Richter scale, resulting in extensive devastation across 11 provinces. According to data provided by the World Health Organization, the earthquakes resulted in a death toll of 51,000 and affected 9.1 million people, causing the displacement of 3 million individuals and the provision of accommodation for over 3 million people. The region experienced numerous subsequent aftershocks. The aftermath saw the collapse or severe damage of no fewer than 298,000 buildings. Earthquakes represent a well-explored phenomenon. The devastating impact of these seismic events goes beyond mere physical destruction and loss of life; it extends to people's aspirations and future plans, causing disruptions to the natural trajectory of their lives. While the anguish experienced by those who've lost loved ones cannot be alleviated, and the reality of the disaster cannot be undone, there may be measures we can adopt to alleviate its repercussions. A fundamental protective element, psychological flexibility, emerges as a means to mitigate the adverse aftermath of earthquakes. This trait empowers individuals to embrace psychological liberation by acknowledging their present circumstances and openly investigating the facets that are within and beyond their control. Natural calamities possess the capacity to reshape our perspective on the world. One's outlook on the future, self-perception, and perception of others undergo transformation compared to our pre-earthquake mindset. The seismic event disrupts the innate cognitive flow, triggering introspection about personal safety, one's role in the world, and the significance underlying social connections. The once-steadfast sense of security is replaced by a belief that danger looms, with vulnerability a constant companion. Traditional cognitive-behavioral therapy (CBT) often challenges these fears by demanding evidence-based thinking, while Acceptance and Commitment Therapy (ACT) offers a different approach. Notably, as psychological flexibility increases, so does one's capacity to manage posttraumatic stress symptoms. Self-Help Plus (SH+), an intervention developed by the World Health Organization (WHO), is designed as a stress management program based on the principles of ACT. Although originally intended for group settings, this study adapts the intervention for individual delivery, tailored specifically for adults affected by the earthquakes. SH+ comprises five sessions dedicated to fostering five essential skills: grounding, disengaging from unhelpful thoughts, aligning actions with personal values, practicing kindness, and creating emotional space. While SH+ was originally conceptualized as a group-based intervention designed to foster social support and shared experiences among participants, this study adapts it for a one-on-one format, emphasizing a more personalized therapeutic approach. This individualized intervention is structured to help participants navigate their distress in a targeted, cost-effective, and concise manner. In the context of earthquake survivors, SH+ has the potential to offer a structured, evidence-based method for developing crucial coping skills, even within the individualized delivery model.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for participation in this study, an individual must satisfy all of the following conditions:
* Age 18 years or older
* Have directly experienced the earthquake
* Exhibit elevated levels of psychological distress, indicated by a score exceeding 15 on the Kessler Psychological Distress Scale (K10) (Kessler et al., 2002)
* Display impaired psychosocial functioning, as evidenced by a score surpassing 16 on the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) (WHO, 2010)

Exclusion Criteria:

* An individual meeting any of the subsequent criteria will not be included in this study:
* Presence of acute medical conditions
* Manifestation of imminent suicide risk or demonstration of acute needs/protection risks (assessed with Problem Management Plus (PM+) manual suicidality assessment)
* Affliction with severe mental disorders, such as psychotic disorders or substance dependence (assessed with PM+ manual, observation checklist),
* Experience of severe cognitive impairment, encompassing conditions like severe intellectual disability or dementia (PM+ manual observation checklist)
* Current utilization of mental health care Participants meeting exclusion criteria will be referred for appropriate treatment as required.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Kessler Psychological Distress Scale (K10) | Change from baseline (Before the intervention) to post assessment (1 week and 3 months after the pre-assessment).
  The key parameter of interest will be the extent of psychological distress encountered by the participants, indicated by a score exceeding 15 on the Kessler Psychological Distress Scale (K10). K-10 is a 10-item scale that assesses the psychological distress. Each item is scored from 1 (none of the time) to 5 (all of the time) and ranges between 10 and 50. Higher scores indicate more severe psychological distress.

SECONDARY OUTCOMES:
The Patient Health Questionnaire (PHQ-9) | Change from baseline (Before the intervention) to post assessment (1 week and 3 months after the pre-assessment).
  PHQ-9 is a 9 item questionnaire that measures the severity of depression symptoms. Items are scored as "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score. Higher scores indicate more severe depressive symptoms.
The Generalized Anxiety Disorder Assessment (GAD-7) | Change from baseline (Before the intervention) to post assessment (1 week and 3 months after the pre-assessment).
  GAD-7 is a 7-item measure of general anxiety symptoms that measures anxiety symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day) providing a range between 0 and 21. Higher scores indicate higher levels of anxiety.
The PTSD Checklist for DSM-5 (PCL-5) | Change from baseline (Before the intervention) to post assessment (1 week and 3 months after the pre-assessment).
  The PCL-5 is a 20-item questionnaire that assesses the symptoms of PTSD. Items are scored from 0 (not at all) to 4 (extremely) providing a range between 0 and 16. Higher scores indicate higher levels of PTSD symptoms.
The Prolonged Grief Disorder Assessment (PG-13) | Change from baseline (Before the intervention) to post assessment (1 week and 3 months after the pre-assessment).
  The PG-13 is a 13-item scale that assesses prolonged grief disorder. For items 1, 2, 4, and 5, respondents provide ratings on a frequency scale, with options ranging from "not at all" to "several times a day," scored from 1 to 5. Items 6 to 12, on the other hand, are assessed on an intensity scale, where respondents rate from "not at all" to "overwhelmingly," also scored from 1 to 5.
Psychological Flexibility Scale | Change from baseline (Before the intervention) to post assessment (1 week and 3 months after the pre-assessment).
  Psychological Flexibility Scale is a 28-item scale that measures psychological flexibility. Each item is scored from 1 (not at all) to 7 (all of the time). The lowest score that can be obtained from the scale is 28, while the highest score is 196. High scores from each subscale in the scale's items reflect high psychological flexibility.
WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | Change from baseline (Before the intervention) to post assessment (1 week and 3 months after the pre-assessment).
  WHODAS is a 12-item scale that assesses ability to engage in daily activities. Each item is scored from 0 (none) to 4 (extreme) and ranges between 0 and 48. Higher scores indicate more daily dysfunctioning.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Acarturk, P.h.D, Principal Investigator — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tol WA, Augustinavicius J, Carswell K, Brown FL, Adaku A, Leku MR, Garcia-Moreno C, Ventevogel P, White RG, van Ommeren M. Translation, adaptation, and pilot of a guided self-help intervention to reduce psychological distress in South Sudanese refugees in Uganda. Glob Ment Health (Camb). 2018 Jul 27;5:e25. doi: 10.1017/gmh.2018.14. eCollection 2018. PMID 30128161